CLINICAL TRIAL: NCT01383512
Title: Medical and Economical Evaluation of Upper Limb's Rehabilitation Robotics After a Stroke
Brief Title: Rehabilitation Robotics After a Stroke
Acronym: REM_AVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REM_AVC
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Subacute Stroke
Keywords: stroke; rehabilitation; robotics; motor control; upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rehabilitation robotics (Experimental): Subjects will be practicing an Armeo Spring rehabilitation program in addition to their usual care (1.5h/day,5d/week) 1h/day 5d/week 4 weeks.
  Interventions: Device: ARMEO Spring
- Self-rehabilitation (Active Comparator): Subject will associated to there classical care 1 hours, 5 days per week during 4 weeks, of self rehabilitation.
  Interventions: Other: Self rehabilitation
- Healthy volunteer (Other): 20 healthy volunteer will be recruiting and using ARMEO Spring. All volunteer will repeat 5 times the same program on the medical device.
  Interventions: Device: ARMEO Spring

INTERVENTIONS:
Device: ARMEO Spring — Use of the device 1 hour per day, 5 days per week during 4 weeks
  Arms: Healthy volunteer; Rehabilitation robotics
Other: Self rehabilitation — Subject have to realised alone rehabilitation exercises 1 hour per day, 5 days per week during 4 weeks.
  Arms: Self-rehabilitation

SUMMARY:
Upper limb motor control after a stroke may be improved with rehabilitation robotics at a subacute stage. The aim of this multicenter controled randomized single blind study is to define the place of rehabilitation robotics at this phase of the rehabilitation process. Both groups will realize the same time of rehabilitation. The cost benefit ratio will be compared in each group through medical assessment of improvement and definition of the costs due to the rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke of the middle cerebral arteria territory
* 18 to 80 years old
* stroke onset between 3 weeks to 3 months,with or without aphasia, with or without lateral neglect and homonymous hemianopia, with or without visual neglect
* 10<or= Fugl Meyer upper limb Score <or= 40
* upper limbs pain less or equal than 3/10 (VAS)
* inpatient or outpatient rehabilitation
* signed inform consent

Exclusion Criteria:

* ischemic or hemorrhagic stroke of anterior or posterior cerebral artery
* ischemic or hemorrhagic stroke of the brainstem
* major aphasia evaluated by a Boston Diagnostic Aphasia Examination (BDAE) score less or equal to 3
* asthenia not allowing to work 60 minutes with the robot.
* serious visual deficiency not allowing to use the robot
* impossibility to install the arm on the robot because of a serious and uncontrolled spasticity or for any other reason
* pronounced and constant muscular contractures, or deformation affecting the use of the extremity
* upper limb's pain superior to 3/10 and/or being worse at the active and passive mobilization
* serious infection and/or instability of vital functions
* perfusion of the affected upper limb not removable
* incapacity to stay on a chair
* contraindicated sitting position
* permanent deviation of the head and\or of the eyes
* perturbed or non-cooperative patient
* patients that must have to be isolated due to an infection process
* bone fracture of the paretic limb with an onset less than 3 months stabilized or not

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer upper limb motor score | Day 30
  Increase of the Fugl Meyer score between day 0 and day 30 with a difference between groups by at least 4 points

SECONDARY OUTCOMES:
Costs | One year
  The rehabilitation costs will be assessed for each group through medical and physiotherapist consultations, hospitalization costs, day of return to work if concerned.
Stroke impact scale (SIS) | One year
  The quality of life will be assessed through the SIS.
Visual analog scale (VAS) | Day 7,14,21,30, 90,180, 360
  The pain of the shoulder and the upper limb will be assessed in different positions
Modification of motor control | Day 30
  Parameter and result of rehabilitation program on ARMEO spring are saved. Data of patient in rehabilitation robotics and healthy volunteer arms will be compared in order to evaluate the modification of the motor control at Day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier REMY-NERIS, Professor, Principal Investigator — University Hospital, Brest
Locations (23):
- France (23):
  - CHU d'Amiens, Amiens
  - CRRRF, Angers
  - CHU de Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - Centre Bouffard Vercelli, Cervera de la Marenda
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CH de Garches, Garches
  - EMPR Le Normandy, Granville
  - CHU de Nîmes, Le Grau-du-Roi
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Lyon, Lyon
  - CRF de Valmante, Marseille
  - CHU de Montpellier, Montpellier
  - IRR de Nancy, Nancy
  - CHU de Nantes, Nantes
  - APHP - Hôpital La Salpétriere, Paris
  - APHP - Hôpital Lariboisière, Paris
  - CMRRF Kerpape, Ploemeur
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Cornec G, Lempereur M, Mensah-Gourmel J, Robertson J, Miramand L, Medee B, Bellaiche S, Gross R, Gracies JM, Remy-Neris O, Bayle N. Measurement properties of movement smoothness metrics for upper limb reaching movements in people with moderate to severe subacute stroke. J Neuroeng Rehabil. 2024 May 29;21(1):90. doi: 10.1186/s12984-024-01382-1. PMID 38812037
- [Derived] Remy-Neris O, Le Jeannic A, Dion A, Medee B, Nowak E, Poiroux E, Durand-Zaleski I; REM Investigative Team*. Additional, Mechanized Upper Limb Self-Rehabilitation in Patients With Subacute Stroke: The REM-AVC Randomized Trial. Stroke. 2021 Jun;52(6):1938-1947. doi: 10.1161/STROKEAHA.120.032545. Epub 2021 Apr 29. PMID 33910364